CLINICAL TRIAL: NCT04879576
Title: The Effects of Telerehabilitation on Respiratory Functions, Quality of Life, Exercise Capacity, Fatigue and Psychosocial Factors in Patients With COPD
Brief Title: The Effects of Telerehabilitation in Patients With COPD
Acronym: COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Beyza Karakaş, Student, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KKUniversity
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: COPD
Keywords: Telerehabilitation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Therapeutics; Telerehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental)
  Interventions: Other: Treatment
- Control Group (No Intervention)

INTERVENTIONS:
Other: Treatment — Telerehabilitation including pulmonary rehabilitation and posture exercises at 8 weeks in total with 2 sessions per week
  Other Names: telerehabilitation
  Arms: Treatment Group

SUMMARY:
Chronic Obstructive Pulmonary Disease is a serious public health problem worldwide and it is a leading cause of mortality and morbidity. Nowadays, COPD patients are increasing in all societies and the problems that arise during the life of these patients increase the need for care and rehabilitation. Pulmonary rehabilitation has proven to be the best supportive treatment for individuals with COPD. However, there are difficulties in rehabilitation practices in terms of the fragility of patients, transportation and access problems. Telerehabilitation allows patients who cannot access rehabilitation due to their geographical, economic or physical disabilities to benefit from rehabilitation services. There are different studies demonstrating the effect of telerehabilitation in COPD patients and confirming that it is safe, but it is a developing area and has a limited area of use.

In this randomized controlled study, it is aimed to examine the effect of telerehabilitation training on respiratory functions, exercise capacity, quality of life, fatigue and psychosocial factors in individuals with COPD via video conferencing including respiratory exercises and postural exercises.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with chronic obstructive pulmonary disease according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria
* Not having an attack in the last 2 months
* Volunteering to participate in the study
* Being between the ages of 40-80
* To have a device that can be used in telerehabilitation application and an active internet connection.

Exclusion Criteria:

* Unstable angina, previous myocardial infarction, severe congestive heart failure resistant to medical therapy, uncontrolled hypertension, cancer, neurological or musculoskeletal disorders with functional limitations
* Currently addicted to alcohol or drugs
* Having an injury to the lower extremity such as sprains, sprains or fractures in the last 6 months, not being able to perform independent ambulation
* Having serious vision and hearing problems
* Having severe cognitive impairment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in respiratory functions on the spirometry at week 8 | Baseline - Week 8
  Spirometry is a standard test doctors use to measure how well your lungs are functioning. The test works by measuring airflow into and out of your lungs.Spirometry measures two key factors: expiratory forced vital capacity (FVC) and forced expiratory volume in one second (FEV1).
Change from Baseline in exercise capacity on six-minute walk test at week 8 | Baseline - Week 8
  The six-minute walk test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.A lower score (reflecting less distance covered in 6 minutes) indicates worse function.
Change from Baseline in health-related quality of life on Saint George's Respiratory Questionnaire at week 8 | Baseline - Week 8
  Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease.Scores range from 0 to 100, with higher scores indicating more limitations.
Change from Baseline in psychosocial factors on Beck Depression and Beck Anxiety Inventory at week 8 | Baseline - Week 8
  Beck Depression Inventory is a self-assessment scale that determines the risk of individuals in terms of depression and measures the level of depressive symptoms and the change in severity.Beck Anxiety Inventory is a likert type self-assessment scale that determines the frequency of anxiety symptoms experienced by individuals. The high score the individual gets from the scale indicates the severity of anxiety experienced.
Change from Baseline in fatigue on COPD and Asthma Fatigue Scale at week 8 | Baseline - Week 8
  The COPD and Asthma Fatigue Scale , was developed for use in clinical trials and other studies in respiratory diseases. The COPD and Asthma Fatigue Scale was intended to be sufficiently comprehensive to capture fatigue experienced by patients with either asthma or COPD, yet be brief and patient centered.

SECONDARY OUTCOMES:
Change from Baseline in dyspnea on Modified Medical Research Council Dyspnea Scale at week 8 | Baseline - Week 8
  The modified Medical Research Council (mMRC) scale is the most commonly used validated scale to assess dyspnea in daily living in chronic respiratory diseases. It is a scale scored between 0 and 5 based on various factors causing dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Beyza Karakaş, Study Director — Graduate student at Kırıkkale University; Meral Sertel, Study Chair — Associate professor at Kırıkkale University; Selma Demir, Principal Investigator — Chest Diseases Specialist at Kırıkkale High Specialization Hospital
Locations (1):
- Kırıkkale High Specialization Hospital, Kırıkkale, Turkey (Türkiye)

REFERENCES:
- [Derived] Avci B, Sertel M, Demir S. The effect of posture and breathing exercises applied with telerehabilitation on respiratory functions, exercise capacity, fatigue, and psychosocial factors in chronic obstructive pulmonary disease patients. J Bodyw Mov Ther. 2025 Dec;45:953-961. doi: 10.1016/j.jbmt.2025.09.046. Epub 2025 Oct 16. PMID 41316669